CLINICAL TRIAL: NCT02118285
Title: Indoleamine-2,3-dioxygenase (IDO) Inhibition With INCB024360 and Intraperitoneal Delivery of Allogeneic Natural Killer Cells for Women With Recurrent Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: Intraperitoneal Natural Killer Cells and INCB024360 for Recurrent Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012LS101; MT2013-11 (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2014-03-26; First posted 2014-04-21 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
Keywords: Ovarian cancer; Fallopian cancer; Primary peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; IL32 protein, human; Interleukin-2; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Haploidentical donor NK cells and IL-2 are infused intraperitoneally (IP) after a non-myeloablative preparative regimen of cyclophosphamide and fludarabine. INCB024360, at the assigned dose, begins 2 days before the NK cell infusion and continues twice daily for 90 days.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: NK cells; Biological: IL-2; Drug: INCB024360

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 25 mg/m^2 IV on days -6 through -2 from NK cell infusion
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide 30 mg/kg IV on days -5 and -4 from NK cell infusion
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune
Biological: NK cells — CD3-/CD19- selected NK cells administered by intraperitoneal (IP) infusion on day 0
  Other Names: Natural Killer Cells
Biological: IL-2 — IL-2 at 6 million units/dose IP 3 times a week x 6 doses with the 1st dose given immediately after the NK cell infusion
  Other Names: Interleukin 2
Drug: INCB024360 — INCB024360 at assigned dose by mouth twice a day begin day -2 and continue for 90 days (+/- 3 days)

SUMMARY:
This is a single center phase I trial designed to determine the maximum tolerated dose (MTD) of the oral IDO inhibitor INCB024360 when administered as part of a larger regimen of intraperitoneal (IP) delivery of haploidentical donor NK cells and IL-2 after a non-myeloablative cyclophosphamide/fludarabine (Cy/Flu) preparative regimen for the treatment of recurrent ovarian, fallopian tube, and primary peritoneal cancer.

DETAILED DESCRIPTION:
Haploidentical donor NK cells and the 1st dose of IL-2 are infused intraperitoneally (IP) after a non-myeloablative preparative regimen of cyclophosphamide and fludarabine. IP IL-2 continues three times a week for 5 additional doses. INCB024360, at the assigned dose, begins 2 days before the NK cell infusion (on day -2) and continues twice daily for 90 days.

Follow-up for disease response and survival is for 1 year from the NK cell infusion with the possibility of re-treatment for patients who experience at least a clinical benefit for a minimum of 6 months prior to disease progression.

The MTD of INCB024360 will be determined using the continual reassessment method (CRM). The 1st 2 patients will be enrolled at dose level 1 (50 mg bid) of INCB024360. Each new cohort of 2 patients will be sequentially assigned to most appropriate dose by the study statistician based on the updated toxicity profile. Up to 4 dose levels of INCB024360 will be tested (50, 100, 200, and 300 mg bid) with a dose level -1 (25 mg bid) used in the event that 50 mg bid proves to be too toxic. The MTD will be identified when the total sample size of 20 patients is exhausted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer that has failed or progressed after at least 1 prior salvage chemotherapy regimen directed at recurrent/metastatic disease.
* Measurable disease per disease specific RECIST version 1.1- patients with bone as their only site of disease will not be eligible
* If history of brain metastases must be stable for at least 3 months after treatment - A brain CT scan will only be required in subjects with known brain metastases at the time of enrollment or in subjects with clinical signs or symptoms suggestive of brain metastases.
* Available related HLA-haploidentical NK cell donor by at least Class I serologic typing at the A&B locus
* Age 18 years or older
* GOG Performance Status ≥ 2 - refer to appendix III
* Adequate organ function as determined by the following criteria within 14 days of the start of the preparative regimen, unless otherwise noted:

  * Bone marrow: platelets ≥ 80,000 x 109/L and hemoglobin ≥ 9 g/dL, unsupported by transfusions; absolute neutrophil count (ANC) ≥ 1000 x 109/L, unsupported by G-CSF or granulocytes
  * Renal function: estimated glomerular filtration rate (GFR) of ≥ 50 ml/min (based on the Fairview Laboratories formula at time of screening)
  * Liver function: total bilirubin < 1.5 times upper limit of institutional normal; AST, ALT, and alkaline phosphatase < 3 times upper limit of institutional normal
  * Cardiac: Left ventricular ejection fraction > 40% (within 28 days of treatment start)
  * Pulmonary function: > 50% corrected DLCO and FEV1, if presence of pleural effusion due to metastatic disease > 40% corrected DLCO and FEV1 is acceptable (within 28 days of treatment start)
* Able to be off prednisone or other immunosuppressive medications other than that prescribed per protocol for at least 3 days prior to Day 0
* At least 14 days must lapse between last prior anti-cancer treatment and 1st day of preparative regimen
* Not pregnant or lactating - The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. Participants of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy and agree to use adequate birth control during study treatment.
* Able to tolerate intraperitoneal (IP) port placement and IP treatment administration in the opinion of the enrolling investigator
* Voluntary written consent

Exclusion Criteria:

* Active infection - must be afebrile and off antibiotics
* Receiving monoamine oxidase inhibitors (MAOI)s or drug which as significant MAOI activity (meperidine, linezolid, methylene blue) within 21 days of 1st dose of fludarabine
* Requiring potent CYP3A4 inducers or inhibitors
* Have ever had Serotonin Syndrome after receiving one or more serotonergic drugs
* Prior therapy with anti-CTLA-4 antibody, anti PD-1, or an experimental immune system-targeted therapy
* Use of any UGT1A9 inhibitor including: diclofenac, imipramine, ketoconazole, mefenamic acid, and probenecid from screening through follow-up period.
* Undergone an organ transplant(s) including allogeneic stem cell or bone marrow transplants.
* Unstable cardiovascular disease (eg, uncontrolled hypertension, peripheral vascular disease, congestive heart failure, cardiac arrhythmia, or acute coronary syndrome) within 6 months of starting study treatment.
* Any gastrointestinal condition causing malabsorption or obstruction (eg, celiac sprue, gastric bypass surgery, strictures, adhesions, history of small bowel resection, blind loop syndrome). Unable or unwilling to swallow tablets BID.
* Active autoimmune process (eg rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease, etc.) or who have been receiving therapy for an autoimmune or inflammatory disease. Vitiligo, thyroiditis, or eczema is permitted if patient is otherwise eligible
* Known HIV-positivity
* History of hepatitis or positive serology as follows:

  * Hepatitis B (HepB) screening testing required:
* HepB SAg (hepatitis B surface antigen);
* Anti-HepB SAg (antibody against hepatitis B surface antigen);
* Anti-Hepatitis B core IgG (antibody against hepatitis B core antigen).
* Hepatitis B core IgM antibody

  * Hepatitis C screening testing required:
* HCV-antibody (antibody against hepatitis C virus);
* HCV-RNA (serum test for circulating virus, based on detecting RNA)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-07-28 (Actual); Primary Completion 2015-11-12 (Actual); Study Completion 2015-11-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of INCB024360 | 90 days
  To determine the maximum tolerated dose (MTD) of INCB024360 when administered with intraperitoneal haploidentical donor NK cells/IL-2 after a nonmyeloablative cyclophosphamide/fludarabine (Cy/Flu) preparative regimen in patients with recurrent ovarian, fallopian tube, and primary peritoneal cancer

SECONDARY OUTCOMES:
Initial tumor response | 90 days
  The proportion of patients with initial tumor response (CR or PR)
Duration of tumor response | 1 year
  Duration of tumor response
Progression-free survival | 5 years
  Average time to progression.
Overall survival | 5 years
  Average length of survival after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Geller, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States